CLINICAL TRIAL: NCT03760666
Title: A Phase 1b/2a Open-label, Multi-center Study to Assess the Safety, Efficacy and Pharmacokinetics of Intrapatient Dose-adjusted Brequinar and Inhibition of Dihydroorotate Dehydrogenase (DHODH) in Adult Subjects With AML
Brief Title: A Study of Brequinar in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No efficacy observed, COVID-19 caused sites to shut down
Sponsor: Clear Creek Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCB-01
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: DHODH; Brequinar; Differentiation; IMPDH Inhibition
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — brequinar; Ribavirin

STUDY DESIGN:
Intervention Model Description: Subjects start dosing with brequinar alone; Cohort 2 subjects may roll over into ribavirin dosing; Cohort 3 subjects started with brequinar monotherapy then added ribavirin dosing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brequinar/Brequinar + Ribavirin (Experimental): Brequinar and ribavirin were dosed orally; brequinar starting doses ranged from 200 mg/m2 to 500 mg/m2. Brequinar doses were adjusted by cohort for starting dose and regimen (either twice-weekly or once-weekly). In addition, the dose for each participant was also adjusted (either escalated or decreased) based on safety, brequinar PK and levels of dihydroorotate (DHO). Ribavirin 1000 mg twice a day (bid) was added in combination with brequinar for the final 3 study participants.
  Interventions: Drug: Brequinar/Brequinar + Ribavirin

INTERVENTIONS:
Drug: Brequinar/Brequinar + Ribavirin — The first 14 participants had brequinar monotherapy; the final 3 subjects were also exposed to a combination of brequinar + ribavirin.

SUMMARY:
A Phase 1b/2a multi-center, open-label, non-randomized study to assess the safety, tolerability and efficacy of dose-adjusted brequinar in adult subjects with acute myeloid leukemia (AML). Ribavirin BID may be added to brequinar twice weekly in eligible subjects.

DETAILED DESCRIPTION:
Up to 27 subjects will be entered in this Phase 1b/2a multi-center, open-label, non-randomized study to assess the safety, tolerability and efficacy of dose-adjusted brequinar in adult subjects with acute myeloid leukemia (AML). Active Cohort 2 subjects on brequinar alone twice weekly may roll over into brequinar twice weekly + ribavirin BID. Cohort 3 subjects will begin treatment with brequinar alone twice weekly then move to brequinar twice weekly + ribavirin BID as tolerated. Both the brequinar and ribavirin doses may be adjusted based on safety, tolerability, and enzyme inhibition levels.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Willing and able to provide written informed consent for the trial.
2. Patients 18 years of age or older, with relapsed/refractory AML by World Health Organization classification, T-cell leukemia (T-ALL), bi-lineal leukemia (BLL), or mixed phenotypic acute leukemia (MPAL) and who have exhausted available therapy.
3. ECOG Performance Status 0 to 2.
4. 12-lead ECG with no clinically unacceptable findings; adequate cardiac function/NYHA Class 0 to 2.
5. Adequate hepatic function (unless deemed to be related to underlying leukemia).

   1. Direct bilirubin ≤ 2 x ULN
   2. ALT ≤ 3 x ULN
   3. AST ≤ 3 x ULN
6. Adequate renal function as documented by creatinine clearance ≥ 50 mL/min based on the Cockcroft-Gault equation.
7. In the absence of rapidly proliferative disease, the interval from prior leukemia-directed therapy to first dose of study drug will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy) agents. Use of supportive care measures per institution's standard of care is permitted at any time.
8. The effects of brequinar on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 90 days after completion of brequinar administration.
9. Male subjects must agree to refrain from sperm donation from initial study drug administration until 90 days after the last dose of study drug.

Exclusion Criteria:

1. Patients in need of immediate leukapheresis.
2. Any concurrent uncontrolled clinically significant medical condition, laboratory abnormality, or psychiatric illness that could place the participant at unacceptable risk of study treatment.
3. QTc interval using Fridericia's formula (QTcF) ≥ 470 msec. Participants with a bundle branch block and prolonged QTc interval may be eligible after discussion with the medical monitor.
4. Pre-existing liver disease.
5. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions:

   a. Intrathecal chemotherapy for prophylactic use or maintenance of controlled CNS leukemia.
6. Presence of graft versus host disease (GVHD) which requires an equivalent dose of ≥ 0.5 mg/kg/day of prednisone or therapy beyond systemic corticosteroids (e.g. cyclosporine or other calcineurin inhibitors or other immunosuppressive agents used for GVHD).
7. Active cerebrospinal involvement of AML, T-cell leukemia (T-ALL), bi-lineal leukemia (BLL), or mixed phenotypic acute leukemia (MPAL).
8. Diagnosis of acute promyelocytic leukemia (APL)
9. Clinically active hepatitis B (HBV) or hepatitis C (HCV) infection.
10. Severe gastrointestinal or metabolic condition that could interfere with the absorption of oral study medication.
11. Prior malignancy, unless it has not been active or has remained stable for at least 2 years. Participants with treated non-melanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible if definitive treatment for the condition has been completed. Participants with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if at the active surveillance stage, hormonal therapy has been initiated, or the malignancy has been surgically removed or treated with definitive radiotherapy.
12. Nursing women or women of childbearing potential (WOCBP) with a positive pregnancy test.
13. Documented hemoglobinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Clear Creek Bio is committed to responsible data sharing regarding the clinical trials we sponsor. Data that may be shared include access to anonymized participant and trial level data (analysis data sets), as well as other information (e.g., protocol) as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Requests for data can be submitted at any time and if the below conditions are met data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Requests for data may be made by qualified researchers who plan to engage in rigorous, independent scientific research. Data will be provided following review and approval of a research proposal including a formal statistical analysis plan and execution of a Data Sharing Agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1 (N = 5) 12/20/2018 - 04/01/2019. Cohort 2 (N = 11) 10/25/2019 - 11/20/2020. Cohort 3 (N = 1) 01/12/21 - 02/03/2021. Participants were enrolled at hematology oncology units at major hospitals. Only 17 of the 27 planned participants were enrolled due to lack of efficacy with either brequinar monotherapy or the brequinar + ribavirin combination. Participants were to be treated in the study for up to one year.
Pre-assignment Details: All subjects had relapsed/refractory AML and had no other viable treatment options. Data were reported and analyzed by cohort.
Groups:
- Cohort 1: 5 subjects were enrolled in this cohort and started dosing at 500 mg/m2 twice weekly
- Cohort 2: Six (6) Cohort 2 subjects started dosing with brequinar monotherapy at 500 mg/m2 on a once-weekly basis and five (5) Cohort 2 subjects started dosing with brequinar monotherapy at 350 mg/m2 on a once-weekly basis.
- Cohort 3: One subject was enrolled into this cohort and started dosing with brequinar monotherapy at 350 mg/m2 on a once-weekly basis. Ribavirin was added at 1000 mg p.o. BID.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 5 | 11 | 1
Completed | 0 | 0 | 0
Not Completed | 5 | 11 | 1
Not completed — Adverse Event | 2 | 4 | 1
Not completed — AML Disease Progression | 3 | 3 | 0
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data were reported and analyzed by cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 5 | 11 | 1 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (20.89) | 72.5 (7.13) | 66.0 (0) | 68.8 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 5 | 8 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 10 | 1 | 13
  Unknown or Not Reported | 3 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 6 | 1 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 11 | 1 | 17
Body Surface Area [Mean (Standard Deviation); unit: meters squared] | 1.94 (0.126) | 1.82 (0.306) | 2.0 (0) | 1.86 (0.259)
ECOG (European Cooperative Oncology Group [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working). The range is 0 to 5; A score of 0 indicates fully active without restrictions, a score of 5 is Dead.
  Participants
    ECOG Score of 0 | 2 | 1 | 0 | 3
    ECOG Score of 1 | 2 | 9 | 0 | 11
    ECOG Score of 2 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: The number of participants with grade 3 or greater treatment-related adverse events as assessed by CTCAE v. 4.03.
Time Frame: 12 months
Population: The Safety Population was used for this analysis. The Safety Population consisted of all subjects who were enrolled in the study and received at least one dose of brequinar. Data were reported and analyzed by cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: The 5 subjects in Cohort 1 started dosing with brequinar monotherapy at 500 mg/m2 on a twice-weekly basis.
- Cohort 2: A total of 11 subjects were enrolled into Cohort 2. Six (6) Cohort 2 subjects started dosing with brequinar monotherapy at 500 mg/m2 on a once-weekly basis and five (5) Cohort 2 subjects started dosing with brequinar monotherapy at 350 mg/m2 on a once-weekly basis.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 11 | 1
Participants | 2 | 3 | 1

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The number of participants in the Efficacy Analysis Set with best overall response of one of the responses of CR, CRi, CRh, PR, of MLFS. No participant met the efficacy endpoint to be included in this analysis
Time Frame: 12 months
Population: The Efficacy Analysis Set was a subset of the Safety population with measurable AML disease at baseline and at least one post-baseline disease response assessment. No subjects achieved this status. Data were reported and analyzed by cohort.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Complete Remission (CR) Rate
Description: The proportion of subjects in the Efficacy Analysis Set with best overall response of CR. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Complete Remission With Incomplete Hematologic Recovery (CRi) Rate
Description: The proportion of subjects in the Efficacy Analysis Set with a best overall response of CRi. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Complete Remission With Partial Hematological Recovery (CRh) Rate
Description: The proportion of subjects in the Efficacy Analysis Set with a best overall response of CRh. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Groups:
- Cohort 1: All subjects started dosing with brequinar monotherapy at 500 mg/m2 on a twice-weekly basis.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Morphologic Leukemia Free State (MLFS) Rate
Description: The proportion of subjects in the Efficacy Analysis Set with a best overall response of MLFS. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Partial Remission (PR) Rate
Description: The proportion of subjects in the Efficacy Analysis Set with a best overall response of PR. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Event Free Survival (EFS) Rate
Description: Interval between first dose and relapse (>=5% bone marrow blasts, reappearance of blasts in blood, or development of extramedullary disease), disease progression, or both. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: as for outcome 2
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Duration of Response
Description: The duration of response is defined as the number of days from the time response criteria are initially met for CR, CRi, CRh, PR, or MLFS (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation. No participant met this efficacy endpoint to be included in this analysis.
Time Frame: Up to approximately 12 months
Population: Subjects with a response. No subjects achieved this status. Data were reported and analyzed by cohort.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Brequinar Pharmacokinetics - Area Under the Curve (AUC)
Description: The plot of drug concentration in blood plasma vs. time.
Time Frame: First day of dosing: baseline (pre-dose), 1 hour, 2 hours, 4 hours, 6 hours.
Population: This population included subjects who completed at least Week 1 of the study. Results are based on Week 1 samples obtained on the first day of dosing at baseline (pre-dose) then at Hour 1, 2, 4, and 6. Data were reported and analyzed by cohort.
Measure: Mean (Standard Deviation); unit: micrograms.hr/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 5 | 11 | 1
micrograms.hr/mL | 501.0 (354.5) | 546.5 (564.1) | 130.5 (0.0)

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: An adverse event is any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
  Events that occur prior to dosing will be entered as medical history; AEs that occur after dosing will be entered on the AE form. Subjects will be questioned and observed for evidence of AEs, whether or not related to study drug.
  Data were reported and analyzed by cohort.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 3/5 | 3/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/5 | 6/11 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 11/11 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=11) | Cohort 3 (N=1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0
Bacteremia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intracranial hematoma (Nervous system disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=11) | Cohort 3 (N=1)
anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 4 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 5 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 0
Tongue erythema (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 0
Fatigue (General disorders) | 1 | 4 | 1
Gait disturbance (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Edema peripheral (General disorders) | 0 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 0
Incision site rash (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 3 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Hemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Nervous system disorders) | 0 | 1 | 0
Depression (Nervous system disorders) | 1 | 0 | 0
Restlessness (Nervous system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0

LIMITATIONS AND CAVEATS:
CCB-01 was a small, open-label study in patients who had exhausted all other therapy options for their relapsed/refractory acute myeloid leukemia (AML). The study was stopped early due to lack of efficacy and inability to recruit new patients during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT03760666/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT03760666/SAP_002.pdf